CLINICAL TRIAL: NCT02719743
Title: An Observer-blind, Dose Ranging Safety and Immunogenicity Study of GSK Biologicals' GSK1557484A Vaccine in Children 6 to Less Than 36 Months of Age
Brief Title: A Dose Ranging Safety and Immunogenicity Study of GlaxoSmithKline (GSK) Biologicals' GSK1557484A Vaccine in Children 6 to Less Than 36 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 116938; 2015-003458-42 (EudraCT Number)
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Influenza
Keywords: children; H5N1; observer-blind; Influenza; dose-ranging
MeSH Terms: conditions — Influenza, Human | interventions — pandemrix

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- H5N1 Formulation 1 Group (Active Comparator): Subjects received 2 primary doses (adjuvanted) at Days 0 and 21 of H5N1 vaccine Formulation 1 and a booster dose (unadjuvanted) at Day 385 of H5N1 vaccine (GSK1557484A). All doses were administered intramuscularly (IM) in anterolateral thigh.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A).
- H5N1 Formulation 2 Group (Experimental): Subjects received 2 primary doses (adjuvanted) at Days 0 and 21 of H5N1 vaccine Formulation 2 and a booster dose (unadjuvanted) at Day 385 of H5N1 vaccine (GSK1557484A). All doses were administered IM in anterolateral thigh.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A).
- H5N1 Formulation 3 Group (Experimental): Subjects received 2 primary doses (adjuvanted) at Days 0 and 21 of H5N1 vaccine Formulation 3 and a booster dose (unadjuvanted) at Day 385 of H5N1 vaccine (GSK1557484A). All doses were administered IM in anterolateral thigh.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A).
- H5N1 Formulation 4 Group (Experimental): Subjects received 2 primary doses (adjuvanted) at Days 0 and 21 of H5N1 vaccine Formulation 4 and a booster dose (unadjuvanted) at Day 385 of H5N1 vaccine (GSK1557484A). All doses were administered IM in anterolateral thigh.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A).
- H5N1 Formulation 5 Group (Experimental): Subjects received 2 primary doses (adjuvanted) at Days 0 and 21 of H5N1 vaccine Formulation 5 and a booster dose (unadjuvanted) at Day 385 of H5N1 vaccine (GSK1557484A). All doses were administered IM in anterolateral thigh.
  Interventions: Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A).

INTERVENTIONS:
Biological: Influenza A (H5N1) Virus monovalent vaccine (GSK1557484A). — All subjects will receive intramuscularly a two-dose primary series (adjuvanted) at a 21 day interval, and a booster dose (unadjuvanted) at Day 385 of GSK1557484A vaccine.

SUMMARY:
The purpose of this study is to assess the safety and immunogenicity of different formulations of GSK Biologicals' influenza candidate vaccine GSK1557484A, in children 6-35 months of age.

DETAILED DESCRIPTION:
Safety and immunogenicity of different formulations administered as a 2-dose schedule in children 6-35 months of age will be evaluated. In addition, the quality of the 2-dose priming will be assessed through the anamnestic response elicited by an antigen challenge (unadjuvanted H5N1) administered 12 months later. The persistence of the immune response approximately 12 months (Day 385) after dose 2 will also be evaluated.

Subjects from each group will be enrolled into the CMI sub-cohort comprising of approximately 100 subjects. Within the participating country(ies), these subjects will be enrolled in only selected/qualified sites.

ELIGIBILITY:
Inclusion Criteria:

* Subject's parent(s)/ Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply with the requirements of the protocol.
* Male or female children 6 months to less than 36 months old at the time of the first vaccination. Children who are not 36 months old as of Day 0, the day of first vaccine dose under this protocol, can be enrolled.
* Written informed consent obtained from the parent(s)/legally acceptable representative(s) [LAR(s)] of the subject prior to performance of any study specific procedure.
* Healthy subjects as established by medical history and standard physical examination before entering into the study.
* Born full-term to be confirmed by interview with parent/LAR or available medical records.

Exclusion Criteria:

* Child in care.
* Medical history of physician-confirmed infection with an H5N1 virus.
* Previous vaccination at any time with an H5N1 vaccine.
* Concurrently participating in another clinical study, or use of an investigational or a non-registered vaccine, pharmaceutical product, or device within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Presence in the parent(s) / LAR(s) of evidence of substance abuse or of neurological or psychiatric diagnoses which, even if stable, are deemed by the investigator to render the parent(s)/LAR(s) unable/unlikely to provide accurate safety reports.
* Acute disease and/or fever at the time of enrolment.
* Administration of immunoglobulins, any blood products, or long-acting immune-modifying drugs during the period starting 3 months before the first dose of study vaccine, or planned administration during the study period.
* History of any neurological disorders or seizures, or Guillain-Barré Syndrome.
* Diagnosed with excessive daytime sleepiness or narcolepsy; or history of narcolepsy in a subject's parent or sibling.
* Administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before the first vaccination.
* Planned administration of any vaccine not foreseen by the study protocol between Day 0 and Day 42 or planned administration of an inactive vaccine within 14 days or of a live attenuated vaccine within 30 days before through 30 days after the booster vaccination. Note: routine vaccinations may be provided on Day 42 after all study assessments have been performed.
* History of any reaction or hypersensitivity likely to be exacerbated by any component of the vaccine; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Any medical condition that in the judgment of the investigator would make intramuscular injection unsafe.
* Chronic administration of immunosuppressants or other immune-modifying drugs during the period starting six months prior to the first vaccine. For corticosteroids, this will mean a dose of prednisone or equivalent of > 2 mg/kg/day of body weight or ≥ 20 mg/day (for persons who weigh ≥ 10 kg). Inhaled and topical steroids are allowed.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Family history of congenital or hereditary immunodeficiency.
* Major congenital defects.
* Any condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 185 (Actual)
Dates: Start 2016-07-07 (Actual); Primary Completion 2018-02-13 (Actual); Study Completion 2018-02-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (5):
- Taiwan (3):
  - GSK Investigational Site, Taichung
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District
- Thailand (2):
  - GSK Investigational Site, Bangkok
  - GSK Investigational Site, Chiang Mai

REFERENCES:
- [Derived] Kim JH, Drame M, Puthanakit T, Chiu NC, Supparatpinyo K, Huang LM, Chiu CH, Chen PY, Hwang KP, Danier J, Friel D, Salaun B, Woo W, Vaughn DW, Innis B, Schuind A. Immunogenicity and Safety of AS03-adjuvanted H5N1 Influenza Vaccine in Children 6-35 Months of Age: Results From a Phase 2, Randomized, Observer-blind, Multicenter, Dose-ranging Study. Pediatr Infect Dis J. 2021 Sep 1;40(9):e333-e339. doi: 10.1097/INF.0000000000003247. PMID 34285165

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Started | 38 | 37 | 38 | 37 | 35
Completed | 37 | 34 | 38 | 36 | 33
Not Completed | 1 | 3 | 0 | 1 | 2
Not completed — Consent withdrawal | 0 | 2 | 0 | 1 | 0
Not completed — Migrated/moved from study area | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group | Total
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35 | 185
Age, Continuous [Mean (Standard Deviation); unit: Months] | 21.9 (8.0) | 22.6 (8.1) | 21.6 (9.2) | 20.8 (8.3) | 20.3 (7.8) | 21.4 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 14 | 16 | 23 | 18 | 88
  Male | 21 | 23 | 22 | 14 | 17 | 97
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian - East Asian Heritage | 21 | 21 | 22 | 21 | 19 | 104
  Asian - South East Asian Heritage | 16 | 16 | 16 | 16 | 16 | 80
  Unspecified | 1 | 0 | 0 | 0 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Humoral Immune Response for A/Indonesia/05/2005 (H5N1) Strain in Terms of Vaccine-homologous Haemagglutination Inhibition (HI) Antibody Titers Following Primary Vaccination
Description: The HI antibody titres were expressed in terms of immunogenicity indices for each group. Immunogenicity index (DGMT) = If the LL of the 95% CI for GMT group ratio is less than 0.25 then DGMT =0. If the LL of the 95% CI for GMT group ratio is greater than 1 then DGMT =1.
Time Frame: At Day 42
Population: Analysis was performed on cohort for analysis of the immunogenicity-fever score which included all subjects who have received all study vaccine dose(s) at Day 42 for whom temperature measurements are available during the first 3 days after both vaccine doses 1 and 2.
Measure: Mean (Full Range); unit: Immunogenicity Index
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Immunogenicity Index | 1 [0 to 1] | 0.54 [0 to 1] | 0.57 [0 to 1] | 0.40 [0 to 1] | 0.34 [0 to 1]

2. Primary Outcome: Humoral Immune Response for A/Indonesia/05/2005 (H5N1) Strain in Terms of Vaccine-homologous Microneutralization (MN) Antibody Titers Following Primary Vaccination
Description: The MN antibody titres were expressed in terms of immunogenicity indices for each group. Immunogenicity index (DGMT) = If the LL of the 95% CI for GMT group ratio is less than 0.25 then DGMT =0. If the LL of the 95% CI for GMT group ratio is greater than 1 then DGMT =1.
Time Frame: At Day 42
Population: Analysis was performed on cohort for analysis of the immunogenicity-fever score which included all subjects who have received all study vaccine dose(s) at Day 42 for whom temperature measurements are available during the first 3 days after both vaccine doses 1 & 2 and with pre & post immune result of antibody of interest.
Measure: Mean (Full Range); unit: Immunogenicity Index
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 31 | 37 | 29 | 35
Immunogenicity Index | 1 [0 to 1] | 0.56 [0 to 1] | 0.57 [0 to 1] | 0.32 [0 to 1] | 0.33 [0 to 1]

3. Primary Outcome: Evaluation of Fever Index for A/Indonesia/05/2005 (H5N1) Strain in Terms of Vaccine-homologous Haemagglutination Inhibition (HI) Antibody Titers Following Primary Vaccination.
Description: Fever index was defined as the average temperature for each vaccine group. Fever index (DR) = The average temperature measurement for each vaccine group. Fever index from Days 0-2 after each dose Any temperature < 38°C (100.4 F) was assigned a value of 0. Any temperature > 40.5°C was assigned a value of 40.5. DR correspond to 243 minus the sum of recorded temperature values for 3 days after (dose 1 and dose 2)/243.
Time Frame: During the 3-day follow-up period (i.e. on the day of vaccination and 2 subsequent days) after Dose 1 and Dose 2.
Population: as for outcome 1
Measure: Mean (Full Range); unit: Degrees Celsius
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Degrees Celsius | 0.84 [0 to 1] | 0.91 [0 to 1] | 0.95 [0 to 1] | 0.93 [0 to 1] | 0.94 [0 to 1]

4. Primary Outcome: Evaluation of Fever Index for A/Indonesia/05/2005 (H5N1) Strain in Terms of Vaccine-homologous Microneutralization (MN) Antibody Titers Following Primary Vaccination.
Description: Fever index was defined as the average temperature for each vaccine group. Fever index (DR)= The average temperature measurement for each vaccine group. Fever index from Days 0-2 after each dose Any temperature < 38°C (100.4 F) was assigned a value of 0. Any temperature > 40.5°C was assigned a value of 40.5. DR correspond to 243 minus the sum of recorded temperature values for 3 days after (dose 1 and dose 2)/243.
Time Frame: During the 3-day follow-up period (i.e. on the day of vaccination and 2 subsequent days) after Dose 1 and Dose 2.
Population: as for outcome 1
Measure: Mean (Full Range); unit: Degrees Celsius
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 31 | 37 | 29 | 35
Degrees Celsius | 0.84 [0 to 1] | 0.91 [0 to 1] | 0.95 [0 to 1] | 0.93 [0 to 1] | 0.94 [0 to 1]

5. Primary Outcome: Mean Geometric Increase (MGI) for Vaccine Homologous and Heterologous HI Antibody Titers Against Each of the Four Vaccine Influenza Strains.
Description: MGI was defined as the geometric mean of the within-subject ratios of the post-vaccination reciprocal HI titer (Day 392) to the pre-vaccination (Day 385) reciprocal HI titer for the vaccine virus. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam/1194/2004 H5N1 (heterologous), Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous) and Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 (heterologous).
Time Frame: At Day 392 (relative to Day 385) post booster vaccination
Population: Analysis was performed on the Adapted According to Protocol (ATP) cohort for immunogenicity which included all vaccinated subjects who had results available for the relevant assay (HI and MN) for all blood samples collected during relevant analysis intervals for ATP-Day 42; ATP-Day 385 (persistence); ATP-Day 392 post booster dose (ATP-booster)
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
Fold change
  Flu A/Indonesia/5/2005 H5N1 HI | 4.9 [3.8 to 6.3] | 6.6 [4.9 to 9.0] | 4.2 [3.4 to 5.3] | 3.6 [2.9 to 4.5] | 3.4 [2.8 to 4.1]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI: number analyzed (Participants) | 33 | 31 | 33 | 31 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI | 5.2 [3.9 to 7.0] | 6.0 [4.2 to 8.5] | 4.0 [3.0 to 5.2] | 3.4 [2.7 to 4.2] | 2.7 [2.3 to 3.3]
  Flu A/Vietnam/1194/2004 H5N1 HI: number analyzed (Participants) | 33 | 31 | 33 | 31 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI | 5.0 [3.7 to 6.8] | 6.3 [4.5 to 8.7] | 3.8 [3.0 to 4.8] | 3.6 [2.9 to 4.5] | 2.8 [2.2 to 3.4]
  Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 HI: number analyzed (Participants) | 33 | 31 | 33 | 31 | 30
  Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 HI | 4.5 [3.2 to 6.5] | 4.9 [3.5 to 6.9] | 3.1 [2.3 to 4.2] | 2.9 [2.2 to 3.8] | 2.4 [2.0 to 3.0]

6. Primary Outcome: Mean Geometric Increase (MGI) for Vaccine Homologous and Heterologous MN Antibody Titers Against Each of the 3 Vaccine Influenza Strains.
Description: MGI was defined as the geometric mean of the within-subject ratios of the post-vaccination (Day 392) reciprocal MN titer to the pre-vaccination (Day 385) reciprocal MN titer for the vaccine virus. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam /1194/2004 H5N (heterologous) and Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous).
Time Frame: At Day 392 (relative to Day 385) post booster vaccination
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
Fold change
  Flu A/Indonesia/5/2005 H5N1 MN | 4.3 [3.3 to 5.7] | 4.8 [3.4 to 6.6] | 3.2 [2.3 to 4.3] | 2.8 [2.0 to 3.8] | 2.5 [2.0 to 3.0]
  Flu A/Vietnam/1194/2004 H5N1 MN: number analyzed (Participants) | 33 | 33 | 35 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN | 2.9 [2.2 to 3.8] | 2.9 [2.1 to 4.1] | 2.9 [2.2 to 3.8] | 2.6 [2.1 to 3.3] | 2.4 [1.9 to 3.1]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN: number analyzed (Participants) | 34 | 33 | 37 | 30 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN | 2.6 [1.9 to 3.5] | 3.0 [2.3 to 4.1] | 2.6 [2.0 to 3.2] | 2.1 [1.6 to 2.8] | 2.8 [2.2 to 3.5]

7. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: Seroconversion rate (SCR) was defined as the proportion of subjects who have either a pre-vaccination reciprocal HI titer less than (<) 10 and a post-vaccination reciprocal titer greater than or equal to (≥) 40, or a pre-vaccination reciprocal HI titer ≥ 10 and at least a 4-fold increase in post vaccination reciprocal titer against the vaccine virus. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam/1194/2004 H5N1 (heterologous), Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous) and Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 (heterologous).
Time Frame: At Days 42, 385 and 392
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Participants
  Flu A/Indonesia/5/2005 H5N1 HI, Day 42 | 36 | 33 | 37 | 31 | 35
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385 | 33 | 26 | 28 | 28 | 21
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392 | 34 | 33 | 37 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42: number analyzed (Participants) | 30 | 24 | 34 | 25 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42 | 30 | 22 | 33 | 23 | 25
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385: number analyzed (Participants) | 31 | 29 | 32 | 25 | 27
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385 | 7 | 6 | 7 | 5 | 6
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392: number analyzed (Participants) | 30 | 29 | 35 | 25 | 27
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392 | 27 | 29 | 26 | 21 | 18
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42: number analyzed (Participants) | 30 | 24 | 34 | 25 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42 | 30 | 22 | 29 | 21 | 24
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385: number analyzed (Participants) | 31 | 29 | 32 | 25 | 27
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385 | 12 | 8 | 9 | 5 | 6
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392: number analyzed (Participants) | 30 | 29 | 35 | 25 | 27
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392 | 29 | 29 | 28 | 22 | 20
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42: number analyzed (Participants) | 30 | 24 | 34 | 25 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42 | 17 | 9 | 10 | 5 | 8
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385: number analyzed (Participants) | 31 | 29 | 32 | 25 | 27
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385 | 1 | 0 | 1 | 0 | 0
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392: number analyzed (Participants) | 30 | 29 | 35 | 25 | 27
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392 | 18 | 15 | 16 | 9 | 6

8. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the 4 Vaccine Influenza Strains.
Description: Seroprotection rate (SPR) was defined as the proportion of subjects with H5N1 reciprocal HI titers ≥ 40 against the tested vaccine virus The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam/1194/2004 H5N1 (heterologous), Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous) and Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 (heterologous).
Time Frame: At Days 0, 42, 385, 392
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Participants
  Flu A/Indonesia/5/2005 H5N1 HI, Day 0 | 0 | 0 | 0 | 0 | 0
  Flu A/Indonesia/5/2005 H5N1 HI, Day 42 | 36 | 33 | 37 | 31 | 35
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385 | 33 | 26 | 28 | 28 | 23
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392 | 34 | 33 | 37 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 0 | 0 | 0 | 0 | 0 | 2
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42 | 32 | 25 | 35 | 28 | 31
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385 | 9 | 8 | 8 | 7 | 6
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392 | 30 | 32 | 27 | 27 | 22
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 0 | 0 | 0 | 0 | 0 | 2
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42 | 32 | 25 | 31 | 26 | 29
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385 | 15 | 10 | 10 | 7 | 8
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392 | 32 | 32 | 29 | 28 | 24
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 0 | 0 | 0 | 0 | 0 | 0
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42 | 19 | 10 | 11 | 7 | 9
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385 | 1 | 1 | 1 | 0 | 1
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392 | 20 | 18 | 16 | 10 | 8

9. Secondary Outcome: Geometric Mean Titers (GMTs) for Humoral Immune Response in Terms of HI Antibodies Against Vaccine-homologous/Heterologous Antigens
Description: GMTs were defined as the geometric mean antibody titres calculated on all subjects post the primary immunization (at Day 0, 42, 385) and 7 days post booster dose (at Day 392). The aggregate variables were calculated for each group. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam/1194/2004 H5N1 (heterologous), Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous) and Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 (heterologous).
Time Frame: At Days 0, 42 and 385 (post the primary immunization), at Day 392 (7 days post booster dose)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Titers
  Flu A/Indonesia/5/2005 H5N1 HI, Day 0 | 5.1 [4.9 to 5.3] | 5.1 [4.9 to 5.3] | 5.1 [4.9 to 5.4] | 5.0 [5.0 to 5.0] | 5.6 [4.9 to 6.5]
  Flu A/Indonesia/5/2005 H5N1 HI, Day 42 | 1118.6 [884.4 to 1414.9] | 858.8 [659.2 to 1118.8] | 913.6 [672.6 to 1241.1] | 640.0 [488.3 to 839.0] | 568.4 [442.7 to 729.8]
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385 | 98.1 [76.7 to 125.4] | 61.5 [47.1 to 80.3] | 72.1 [51.6 to 100.7] | 79.1 [59.2 to 105.6] | 59.6 [45.0 to 79.0]
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392 | 476.2 [348.4 to 650.9] | 407.6 [315.0 to 527.4] | 305.4 [227.1 to 410.6] | 286.2 [216.0 to 379.1] | 201.0 [156.1 to 258.7]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 0 | 5.3 [5.0 to 5.7] | 5.4 [4.8 to 5.9] | 5.3 [5.0 to 5.7] | 5.0 [5.0 to 5.0] | 6.1 [4.9 to 7.6]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42 | 167.1 [128.4 to 217.3] | 135.3 [97.6 to 187.5] | 109.9 [81.2 to 148.7] | 91.5 [70.2 to 119.1] | 78.5 [58.5 to 105.3]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385 | 23.4 [18.8 to 29.2] | 20.8 [16.3 to 26.6] | 17.8 [13.2 to 24.1] | 20.9 [16.1 to 26.9] | 19.5 [14.2 to 26.8]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392 | 125.6 [89.4 to 176.5] | 126.1 [95.2 to 167.0] | 77.6 [54.5 to 110.4] | 70.7 [52.7 to 95.0] | 53.5 [38.6 to 74.2]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 0 | 5.3 [5.0 to 5.7] | 5.0 [5.0 to 5.0] | 5.1 [4.9 to 5.5] | 5.1 [4.9 to 5.4] | 5.8 [4.7 to 7.2]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42 | 128.9 [103.1 to 161.2] | 104.7 [79.0 to 138.6] | 88.9 [63.2 to 125.0] | 77.2 [59.7 to 99.9] | 69.0 [51.7 to 92.0]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385 | 26.0 [20.0 to 33.8] | 21.5 [16.8 to 27.5] | 18.4 [13.2 to 25.7] | 21.3 [16.3 to 27.9] | 20.6 [14.8 to 28.7]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392 | 133.9 [95.5 to 187.7] | 137.5 [107.3 to 176.1] | 76.2 [53.9 to 107.7] | 76.5 [56.8 to 103.1] | 57.8 [41.5 to 80.4]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 0: number analyzed (Participants) | 33 | 30 | 35 | 25 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 0 | 5.3 [4.9 to 5.7] | 5.0 [5.0 to 5.0] | 5.1 [4.9 to 5.3] | 5.2 [4.8 to 5.7] | 5.3 [4.9 to 5.8]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42 | 35.8 [27.9 to 46.0] | 27.8 [21.1 to 36.7] | 22.8 [17.2 to 30.3] | 21.6 [16.7 to 27.8] | 19.9 [15.4 to 25.8]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385 | 9.2 [7.6 to 11.2] | 8.0 [6.4 to 9.9] | 7.4 [6.0 to 9.0] | 7.7 [6.6 to 9.1] | 7.2 [5.8 to 8.8]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392 | 42.6 [29.8 to 60.8] | 37.0 [27.1 to 50.6] | 24.0 [17.1 to 33.6] | 22.6 [16.7 to 30.5] | 17.9 [13.4 to 23.9]

10. Secondary Outcome: Mean Geometric Increase (MGI) for Haemagglutination Inhibition (HI) Antibody Titer Against Each of the 4 Vaccine Influenza Strains
Description: MGI was defined as the geometric mean of the within-subject ratios of the post-vaccination (Day 42) reciprocal HI titer to the pre-vaccination (Day 0) reciprocal HI titer for the vaccine virus. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam/1194/2004 H5N1 (heterologous), Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous) and Flu A/gyrfalcon/Washington/41088-6/2014 H5N8 (heterologous).
Time Frame: At Day 42 (relative to Day 0), at Day 385 (relative to Day 0) and at Day 392 (relative to Day 0)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Fold change
  Flu A/Indonesia/5/2005 H5N1 HI, Day 42 | 219.5 [172.6 to 279.0] | 168.2 [127.4 to 222.0] | 177.7 [131.5 to 240.1] | 128.0 [97.7 to 167.8] | 101.0 [74.8 to 136.4]
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 385 | 19.2 [14.8 to 24.9] | 12.0 [9.2 to 15.8] | 14.0 [10.0 to 19.7] | 15.8 [11.8 to 21.1] | 10.5 [7.6 to 14.5]
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 HI, Day 392 | 93.3 [67.9 to 128.3] | 79.8 [61.5 to 103.5] | 59.4 [44.5 to 79.4] | 57.2 [43.2 to 75.8] | 35.3 [25.9 to 48.1]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 42 | 31.3 [23.5 to 41.6] | 22.9 [17.2 to 30.6] | 20.4 [14.9 to 28.1] | 18.9 [14.0 to 25.5] | 12.6 [9.0 to 17.6]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 385 | 4.2 [3.3 to 5.3] | 3.6 [2.9 to 4.6] | 3.3 [2.4 to 4.5] | 3.9 [2.9 to 5.3] | 3.3 [2.3 to 4.7]
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 HI, Day 392 | 23.4 [16.2 to 33.9] | 22.9 [17.1 to 30.7] | 14.5 [10.1 to 20.7] | 13.9 [9.8 to 19.8] | 9.1 [6.0 to 13.7]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 42 | 24.3 [19.0 to 31.0] | 20.1 [15.2 to 26.7] | 16.7 [11.7 to 23.8] | 15.1 [11.1 to 20.6] | 11.4 [8.4 to 15.6]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 385 | 4.7 [3.5 to 6.2] | 4.1 [3.1 to 5.3] | 3.5 [2.5 to 5.0] | 3.9 [2.8 to 5.4] | 3.6 [2.6 to 5.2]
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 HI, Day 392 | 25.1 [17.3 to 36.4] | 27.1 [20.9 to 35.0] | 14.5 [10.2 to 20.5] | 14.5 [10.0 to 21.1] | 10.1 [6.7 to 15.2]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42: number analyzed (Participants) | 32 | 27 | 36 | 31 | 35
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 42 | 6.7 [5.0 to 9.0] | 5.5 [4.0 to 7.4] | 4.3 [3.2 to 5.8] | 4.1 [3.0 to 5.6] | 3.5 [2.7 to 4.6]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385: number analyzed (Participants) | 34 | 32 | 34 | 31 | 30
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 385 | 1.7 [1.4 to 2.1] | 1.5 [1.2 to 1.8] | 1.4 [1.2 to 1.8] | 1.5 [1.2 to 1.8] | 1.3 [1.1 to 1.6]
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392: number analyzed (Participants) | 33 | 32 | 36 | 31 | 32
  Flu A/gyrfalcon/WA/41088-6/2014 H5N8 HI, Day 392 | 8.1 [5.5 to 12.0] | 7.1 [5.1 to 9.9] | 4.7 [3.3 to 6.7] | 4.2 [3.0 to 6.0] | 3.2 [2.3 to 4.3]

11. Secondary Outcome: Mean Geometric Increase (MGI) for MN Antibodies Against the 3 Vaccine Influenza Strains.
Description: MGI was defined as the geometric mean of the within-subject ratios of the post-vaccination (Day 385) reciprocal MN titer to the pre-vaccination (Day 0) reciprocal MN titer for the vaccine virus. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam /1194/2004 H5N (heterologous) and Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous).
Time Frame: At Day 385 (relative to Day 0)
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Fold change
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 34 | 32 | 37 | 30 | 32
Fold change
  Flu A/Indonesia/5/2005 H5N1 MN: number analyzed (Participants) | 34 | 32 | 37 | 29 | 32
  Flu A/Indonesia/5/2005 H5N1 MN | 17.5 [13.7 to 22.4] | 14.8 [12.6 to 17.5] | 15.3 [12.5 to 18.6] | 17.8 [14.3 to 22.1] | 14.2 [11.8 to 17.1]
  Flu A/Vietnam/1194/2004 H5N1 MN: number analyzed (Participants) | 31 | 32 | 35 | 30 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN | 7.6 [5.5 to 10.3] | 5.8 [4.2 to 8.1] | 5.4 [4.0 to 7.4] | 7.5 [5.8 to 9.8] | 6.1 [4.5 to 8.3]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN: number analyzed (Participants) | 33 | 32 | 37 | 30 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN | 7.0 [5.2 to 9.4] | 5.5 [4.1 to 7.3] | 5.3 [3.8 to 7.3] | 6.9 [5.0 to 9.4] | 4.2 [3.1 to 5.8]

12. Secondary Outcome: Humoral Immune Response for A/Indonesia/05/2005 (H5N1) Strain in Terms of MN Antibodies Against Vaccine-homologous/Heterologous Antigens
Description: MN antibody titers were expressed as Geometric Mean Titers (GMTs). The cut-off of the assay was the seropositivity cut-off of ≥ 1:28. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam /1194/2004 H5N (heterologous) and Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous).
Time Frame: At Days 0, 42, 385 and Day 392
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Titers
  Flu A/Indonesia/5/2005 H5N1 MN, Day 0: number analyzed (Participants) | 36 | 32 | 37 | 29 | 35
  Flu A/Indonesia/5/2005 H5N1 MN, Day 0 | 14.3 [13.7 to 14.8] | 14.0 [14.0 to 14.0] | 14.0 [14.0 to 14.0] | 14.0 [14.0 to 14.0] | 14.0 [14.0 to 14.0]
  Flu A/Indonesia/5/2005 H5N1 MN, Day 42: number analyzed (Participants) | 36 | 32 | 37 | 31 | 35
  Flu A/Indonesia/5/2005 H5N1 MN, Day 42 | 1498.5 [1181.7 to 1900.1] | 1214.3 [921.3 to 1600.6] | 1211.6 [881.3 to 1665.9] | 707.1 [533.1 to 937.9] | 727.4 [545.9 to 969.2]
  Flu A/Indonesia/5/2005 H5N1 MN, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, Day 385 | 250.3 [197.1 to 318.0] | 203.6 [172.8 to 239.8] | 213.8 [175.2 to 260.9] | 247.2 [201.4 to 303.5] | 198.5 [165.1 to 238.7]
  Flu A/Indonesia/5/2005 H5N1 MN, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, Day 392 | 1085.0 [767.5 to 1533.9] | 969.1 [710.1 to 1322.6] | 674.2 [492.3 to 923.3] | 681.0 [496.3 to 934.4] | 489.6 [381.7 to 628.0]
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 0: number analyzed (Participants) | 34 | 32 | 37 | 30 | 35
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 0 | 14.6 [13.8 to 15.4] | 14.6 [13.7 to 15.5] | 14.8 [13.6 to 16.1] | 14.0 [14.0 to 14.0] | 15.2 [13.5 to 17.0]
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 42 | 217.6 [187.7 to 252.2] | 195.2 [156.7 to 243.1] | 177.3 [147.8 to 212.7] | 176.9 [139.0 to 225.2] | 149.3 [117.6 to 189.6]
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 385: number analyzed (Participants) | 33 | 33 | 35 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 385 | 113.0 [85.3 to 149.9] | 88.0 [64.0 to 121.0] | 80.7 [58.7 to 111.1] | 103.6 [80.5 to 133.2] | 89.0 [67.2 to 118.0]
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 392 | 320.0 [259.8 to 394.1] | 256.6 [212.5 to 309.9] | 239.2 [202.5 to 282.7] | 270.4 [237.2 to 308.3] | 216.5 [179.0 to 261.8]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 0: number analyzed (Participants) | 35 | 32 | 37 | 31 | 35
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 0 | 14.6 [13.8 to 15.4] | 14.3 [13.7 to 15.0] | 14.5 [13.5 to 15.7] | 14.6 [13.7 to 15.6] | 15.2 [13.8 to 16.7]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 42 | 179.4 [146.5 to 219.7] | 161.6 [129.4 to 201.9] | 147.1 [116.6 to 185.7] | 161.8 [129.1 to 202.8] | 140.6 [111.8 to 176.8]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 30 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 385 | 102.0 [76.6 to 135.9] | 79.2 [59.3 to 105.8] | 76.3 [55.7 to 104.7] | 100.7 [74.2 to 136.6] | 63.0 [47.0 to 84.4]
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 392 | 262.5 [212.2 to 324.7] | 240.9 [197.7 to 293.6] | 194.8 [157.7 to 240.7] | 202.2 [167.8 to 243.7] | 174.5 [140.5 to 216.8]

13. Secondary Outcome: Vaccine Response Rate (VRR) for Homologous and Heterologous MN Antibodies Against Each of the 3 Vaccine Influenza Strains.
Description: VRR for MN was defined as the incidence rate of subjects with at least a 4-fold increase in post vaccination reciprocal titer relative to pre vaccination titers. The vaccine strains assessed were Flu A/Indonesia/5/2005 H5N1 (homologous), Flu A/Vietnam /1194/2004 H5N (heterologous) and Flu A/duck/Bangladesh/19097/2013 H5N1 (heterologous).
Time Frame: At Day 42, Day 385 (relative to Day 0), Day 392 (relative to Day 0) and D 392 (relative to Day 385)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 33 | 37 | 31 | 35
Participants
  Flu A/Indonesia/5/2005 H5N1 MN, Day 42: number analyzed (Participants) | 36 | 32 | 37 | 29 | 35
  Flu A/Indonesia/5/2005 H5N1 MN, Day 42 | 36 | 31 | 37 | 29 | 35
  Flu A/Indonesia/5/2005 H5N1 MN, Day 385: number analyzed (Participants) | 34 | 33 | 37 | 29 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, Day 385 | 34 | 32 | 37 | 29 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, Day 392: number analyzed (Participants) | 34 | 33 | 37 | 29 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, Day 392 | 34 | 32 | 37 | 29 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, D 392: number analyzed (Participants) | 34 | 33 | 37 | 31 | 32
  Flu A/Indonesia/5/2005 H5N1 MN, D 392 | 21 | 24 | 14 | 15 | 13
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 42: number analyzed (Participants) | 34 | 32 | 37 | 30 | 35
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 42 | 34 | 31 | 36 | 29 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 385: number analyzed (Participants) | 31 | 32 | 35 | 30 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 385 | 27 | 27 | 27 | 28 | 25
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 392: number analyzed (Participants) | 32 | 32 | 37 | 30 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, Day 392 | 31 | 31 | 37 | 30 | 30
  Flu A/Vietnam/1194/2004 H5N1 MN, D 392: number analyzed (Participants) | 33 | 33 | 35 | 31 | 32
  Flu A/Vietnam/1194/2004 H5N1 MN, D 392 | 10 | 10 | 10 | 7 | 6
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 42: number analyzed (Participants) | 35 | 32 | 37 | 31 | 35
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 42 | 34 | 31 | 35 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 385: number analyzed (Participants) | 33 | 32 | 37 | 30 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 385 | 28 | 27 | 29 | 25 | 23
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 392: number analyzed (Participants) | 33 | 32 | 37 | 31 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, Day 392 | 33 | 32 | 36 | 31 | 30
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, D 392: number analyzed (Participants) | 34 | 33 | 37 | 30 | 32
  Flu A/duck/Bangladesh/19097/2013 H5N1 MN, D 392 | 9 | 10 | 8 | 6 | 9

14. Secondary Outcome: Cell Mediated Immunity (CMI) in Terms of T-cell Markers Related to Flu A/Indonesia/05/2005 Antigen.
Description: Antigen-specific CD4+/CD8+ T Cells identified as CD4/CD8+ were analysed for T cells expressing two or more of the following immune markers: CD40 Ligand, Interleukin (IL)-2, Tumor Necrosis Factor alpha (TNF-a), Interferon-gamma (IFN-g). The frequency was presented as number of cytokine-producing CD4+/CD8+ cells per million CD4+/CD8+ cells repsectively. All doubles = T cell expressing at least 2 cytokines.
Time Frame: At Days 0, 42, 385 and 392
Population: Analysis was performed on the Total Vaccinated cohort (CMI sub-cohort) which included all vaccinated subjects for whom data were available. The CMI sub-cohort included approximately 20 vaccinated subjects per group.
Measure: Median (Inter-Quartile Range); unit: cells/million T cells
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 20 | 19 | 19 | 18 | 19
cells/million T cells
  CD4 dble_All (Polypositives), Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD4 dble_All (Polypositives), Day 0 | 55.5 [1.0 to 227.0] | 42.0 [3.0 to 185.0] | 43.0 [1.0 to 90.0] | 89.5 [26.0 to 217.0] | 74.0 [1.0 to 277.0]
  CD4 dble_All (Polypositives), Day 42: number analyzed (Participants) | 18 | 19 | 17 | 16 | 16
  CD4 dble_All (Polypositives), Day 42 | 2711.0 [1669.0 to 5165.0] | 1629.0 [707.0 to 4301.0] | 960.0 [432.0 to 1379.0] | 1337.5 [748.0 to 2793.0] | 1372.5 [426.5 to 2911.5]
  CD4 dble_All (Polypositives), Day 385: number analyzed (Participants) | 20 | 18 | 18 | 18 | 17
  CD4 dble_All (Polypositives), Day 385 | 1530.0 [632.5 to 2293.5] | 1255.0 [560.0 to 2096.0] | 1413.0 [469.0 to 1834.0] | 954.0 [495.0 to 1199.0] | 596.0 [373.0 to 1167.0]
  CD4 dble_All (Polypositives), Day 392: number analyzed (Participants) | 20 | 17 | 19 | 18 | 17
  CD4 dble_All (Polypositives), Day 392 | 1417.0 [759.5 to 3955.5] | 1129.0 [582.0 to 3221.0] | 731.0 [448.0 to 1461.0] | 722.5 [260.0 to 907.0] | 832.0 [345.0 to 1497.0]
  CD4 dble_CD40L, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD4 dble_CD40L, Day 0 | 23.0 [1.0 to 56.0] | 19.0 [1.0 to 52.0] | 5.0 [1.0 to 60.0] | 36.0 [1.0 to 85.0] | 26.0 [1.0 to 133.0]
  CD4 dble_CD40L, Day 42: number analyzed (Participants) | 18 | 19 | 17 | 16 | 16
  CD4 dble_CD40L, Day 42 | 1671.0 [635.0 to 3256.0] | 1341.0 [378.0 to 2696.0] | 514.0 [229.0 to 1200.0] | 516.0 [307.5 to 2031.0] | 717.0 [295.5 to 1604.5]
  CD4 dble_CD40L, Day 385: number analyzed (Participants) | 20 | 18 | 18 | 18 | 17
  CD4 dble_CD40L, Day 385 | 1074.0 [562.5 to 2637.0] | 844.0 [425.0 to 1660.0] | 722.0 [323.0 to 1524.0] | 315.0 [148.0 to 511.0] | 588.0 [154.0 to 902.0]
  CD4 dble_CD40L, Day 392: number analyzed (Participants) | 20 | 17 | 19 | 18 | 17
  CD4 dble_CD40L, Day 392 | 1130.5 [801.0 to 3108.5] | 986.0 [340.0 to 1802.0] | 660.0 [213.0 to 1706.0] | 424.0 [239.0 to 645.0] | 325.0 [110.0 to 939.0]
  CD4 dble_IFNγ, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD4 dble_IFNγ, Day 0 | 47.0 [4.0 to 391.0] | 49.0 [1.0 to 352.0] | 24.0 [1.0 to 118.0] | 40.5 [1.0 to 681.0] | 12.0 [1.0 to 259.0]
  CD4 dble_IFNγ, Day 42: number analyzed (Participants) | 18 | 19 | 17 | 16 | 16
  CD4 dble_IFNγ, Day 42 | 803.0 [260.0 to 1627.0] | 406.0 [304.0 to 1481.0] | 266.0 [206.0 to 394.0] | 863.5 [352.5 to 1229.5] | 437.5 [158.5 to 1027.0]
  CD4 dble_IFNγ, Day 385: number analyzed (Participants) | 20 | 18 | 18 | 18 | 17
  CD4 dble_IFNγ, Day 385 | 200.0 [80.0 to 510.0] | 316.5 [70.0 to 569.0] | 248.5 [56.0 to 557.0] | 589.5 [216.0 to 830.0] | 163.0 [62.0 to 355.0]
  CD4 dble_IFNγ, Day 392: number analyzed (Participants) | 20 | 17 | 19 | 18 | 17
  CD4 dble_IFNγ, Day 392 | 459.5 [127.0 to 941.5] | 329.0 [109.0 to 784.0] | 123.0 [74.0 to 465.0] | 423.5 [147.0 to 919.0] | 253.0 [112.0 to 608.0]
  CD4 dble_IL2, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD4 dble_IL2, Day 0 | 89.5 [1.0 to 136.5] | 72.0 [27.0 to 183.0] | 50.0 [1.0 to 76.0] | 47.0 [3.0 to 133.0] | 75.0 [1.0 to 223.0]
  CD4 dble_IL2, Day 42: number analyzed (Participants) | 18 | 19 | 17 | 16 | 16
  CD4 dble_IL2, Day 42 | 3399.5 [1593.0 to 5907.0] | 2438.0 [759.0 to 6212.0] | 1344.0 [508.0 to 1859.0] | 1448.0 [1012.5 to 2993.5] | 1761.5 [577.5 to 3085.5]
  CD4 dble_IL2, Day 385: number analyzed (Participants) | 20 | 18 | 18 | 18 | 17
  CD4 dble_IL2, Day 385 | 1676.5 [779.5 to 2551.5] | 1394.0 [531.0 to 2151.0] | 1366.5 [460.0 to 1938.0] | 870.5 [458.0 to 1223.0] | 621.0 [410.0 to 1556.0]
  CD4 dble_IL2, Day 392: number analyzed (Participants) | 20 | 17 | 19 | 18 | 17
  CD4 dble_IL2, Day 392 | 1502.5 [864.5 to 3500.0] | 1455.0 [672.0 to 3065.0] | 893.0 [627.0 to 1494.0] | 840.0 [192.0 to 1067.0] | 882.0 [338.0 to 1181.0]
  CD4 dble_TNFα, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD4 dble_TNFα, Day 0 | 49.5 [1.0 to 322.0] | 98.0 [1.0 to 249.0] | 62.0 [1.0 to 192.0] | 52.0 [23.0 to 249.0] | 71.0 [29.0 to 296.0]
  CD4 dble_TNFα, Day 42: number analyzed (Participants) | 18 | 19 | 17 | 16 | 16
  CD4 dble_TNFα, Day 42 | 3023.0 [917.0 to 4946.0] | 1970.0 [569.0 to 4382.0] | 840.0 [705.0 to 1446.0] | 1353.0 [723.0 to 2501.0] | 1204.5 [582.5 to 2853.0]
  CD4 dble_TNFα, Day 385: number analyzed (Participants) | 20 | 18 | 18 | 18 | 17
  CD4 dble_TNFα, Day 385 | 1339.0 [765.0 to 2419.5] | 1233.0 [696.0 to 2030.0] | 1277.5 [419.0 to 1921.0] | 1097.5 [547.0 to 1517.0] | 678.0 [463.0 to 1251.0]
  CD4 dble_TNFα, Day 392: number analyzed (Participants) | 20 | 17 | 19 | 18 | 17
  CD4 dble_TNFα, Day 392 | 1743.5 [741.5 to 3863.0] | 1257.0 [504.0 to 2468.0] | 740.0 [394.0 to 1266.0] | 726.5 [433.0 to 1315.0] | 908.0 [620.0 to 1579.0]
  CD8 dble_All (Polypositives), Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD8 dble_All (Polypositives), Day 0 | 3.5 [1.0 to 68.5] | 5.0 [1.0 to 45.0] | 30.0 [1.0 to 40.0] | 47.0 [1.0 to 121.0] | 1.0 [1.0 to 58.0]
  CD8 dble_All (Polypositives), Day 42: number analyzed (Participants) | 17 | 19 | 17 | 16 | 15
  CD8 dble_All (Polypositives), Day 42 | 48.0 [2.0 to 186.0] | 63.0 [42.0 to 238.0] | 45.0 [1.0 to 83.0] | 125.0 [54.5 to 220.5] | 128.0 [10.0 to 323.0]
  CD8 dble_All (Polypositives), Day 385: number analyzed (Participants) | 20 | 18 | 19 | 18 | 17
  CD8 dble_All (Polypositives), Day 385 | 33.5 [1.0 to 108.5] | 62.5 [1.0 to 147.0] | 1.0 [1.0 to 107.0] | 56.0 [1.0 to 194.0] | 1.0 [1.0 to 79.0]
  CD8 dble_All (Polypositives), Day 392: number analyzed (Participants) | 19 | 17 | 19 | 18 | 17
  CD8 dble_All (Polypositives), Day 392 | 63.0 [1.0 to 200.0] | 33.0 [1.0 to 88.0] | 25.0 [1.0 to 70.0] | 60.5 [1.0 to 126.0] | 26.0 [1.0 to 99.0]
  CD8 dble_CD40L, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD8 dble_CD40L, Day 0 | 1.0 [1.0 to 72.5] | 1.0 [1.0 to 21.0] | 1.0 [1.0 to 37.0] | 46.0 [1.0 to 75.0] | 1.0 [1.0 to 57.0]
  CD8 dble_CD40L, Day 42: number analyzed (Participants) | 17 | 19 | 17 | 16 | 15
  CD8 dble_CD40L, Day 42 | 108.0 [7.0 to 147.0] | 25.0 [1.0 to 100.0] | 1.0 [1.0 to 68.0] | 7.5 [1.0 to 60.0] | 83.0 [1.0 to 186.0]
  CD8 dble_CD40L, Day 385: number analyzed (Participants) | 20 | 18 | 19 | 18 | 17
  CD8 dble_CD40L, Day 385 | 88.0 [1.0 to 197.5] | 70.5 [11.0 to 132.0] | 53.0 [1.0 to 93.0] | 4.0 [1.0 to 116.0] | 1.0 [1.0 to 31.0]
  CD8 dble_CD40L, Day 392: number analyzed (Participants) | 19 | 17 | 19 | 18 | 17
  CD8 dble_CD40L, Day 392 | 40.0 [1.0 to 244.0] | 18.0 [1.0 to 95.0] | 14.0 [1.0 to 140.0] | 80.0 [1.0 to 135.0] | 10.0 [1.0 to 55.0]
  CD8 dble_IFNγ, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD8 dble_IFNγ, Day 0 | 41.5 [1.0 to 148.0] | 33.0 [1.0 to 64.0] | 22.0 [1.0 to 53.0] | 78.0 [28.0 to 166.0] | 1.0 [1.0 to 138.0]
  CD8 dble_IFNγ, Day 42: number analyzed (Participants) | 17 | 19 | 17 | 16 | 15
  CD8 dble_IFNγ, Day 42 | 32.0 [1.0 to 129.0] | 77.0 [1.0 to 321.0] | 67.0 [1.0 to 116.0] | 191.5 [60.5 to 329.0] | 131.0 [1.0 to 243.0]
  CD8 dble_IFNγ, Day 385: number analyzed (Participants) | 20 | 18 | 19 | 18 | 17
  CD8 dble_IFNγ, Day 385 | 99.5 [2.5 to 348.0] | 103.0 [1.0 to 322.0] | 31.0 [1.0 to 170.0] | 165.5 [64.0 to 445.0] | 1.0 [1.0 to 251.0]
  CD8 dble_IFNγ, Day 392: number analyzed (Participants) | 19 | 17 | 19 | 18 | 17
  CD8 dble_IFNγ, Day 392 | 52.0 [2.0 to 364.0] | 174.0 [56.0 to 484.0] | 31.0 [1.0 to 206.0] | 119.0 [16.0 to 431.0] | 28.0 [1.0 to 366.0]
  CD8 dble_IL2, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD8 dble_IL2, Day 0 | 1.0 [1.0 to 66.0] | 22.0 [1.0 to 104.0] | 1.0 [1.0 to 49.0] | 1.0 [1.0 to 90.0] | 1.0 [1.0 to 94.0]
  CD8 dble_IL2, Day 42: number analyzed (Participants) | 17 | 19 | 17 | 16 | 15
  CD8 dble_IL2, Day 42 | 1.0 [1.0 to 168.0] | 48.0 [1.0 to 197.0] | 53.0 [1.0 to 166.0] | 65.5 [1.0 to 263.0] | 1.0 [1.0 to 186.0]
  CD8 dble_IL2, Day 385: number analyzed (Participants) | 20 | 18 | 19 | 18 | 17
  CD8 dble_IL2, Day 385 | 1.0 [1.0 to 125.0] | 32.5 [1.0 to 218.0] | 16.0 [1.0 to 111.0] | 14.0 [1.0 to 117.0] | 1.0 [1.0 to 94.0]
  CD8 dble_IL2, Day 392: number analyzed (Participants) | 19 | 17 | 19 | 18 | 17
  CD8 dble_IL2, Day 392 | 63.0 [1.0 to 451.0] | 99.0 [22.0 to 292.0] | 1.0 [1.0 to 70.0] | 64.0 [1.0 to 156.0] | 45.0 [1.0 to 77.0]
  CD8 dble_TNFα, Day 0: number analyzed (Participants) | 20 | 19 | 17 | 18 | 19
  CD8 dble_TNFα, Day 0 | 120.5 [1.0 to 553.0] | 103.0 [1.0 to 516.0] | 34.0 [1.0 to 324.0] | 163.5 [48.0 to 614.0] | 116.0 [1.0 to 521.0]
  CD8 dble_TNFα, Day 42: number analyzed (Participants) | 17 | 19 | 17 | 16 | 15
  CD8 dble_TNFα, Day 42 | 192.0 [52.0 to 485.0] | 396.0 [77.0 to 709.0] | 125.0 [24.0 to 294.0] | 351.5 [153.5 to 970.5] | 756.0 [65.0 to 1557.0]
  CD8 dble_TNFα, Day 385: number analyzed (Participants) | 20 | 18 | 19 | 18 | 17
  CD8 dble_TNFα, Day 385 | 77.5 [15.0 to 477.5] | 366.5 [1.0 to 559.0] | 81.0 [1.0 to 204.0] | 301.5 [29.0 to 641.0] | 212.0 [85.0 to 411.0]
  CD8 dble_TNFα, Day 392: number analyzed (Participants) | 19 | 17 | 19 | 18 | 17
  CD8 dble_TNFα, Day 392 | 217.0 [36.0 to 699.0] | 130.0 [1.0 to 708.0] | 121.0 [26.0 to 238.0] | 310.0 [68.0 to 953.0] | 207.0 [47.0 to 369.0]

15. Secondary Outcome: Number of Subjects Reporting Solicited Local Symptoms
Description: Solicited local AEs assessed were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = cried when limb is moved/spontaneously painful. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after any vaccine dose
Population: Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available.
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Pain, Any | 20 | 15 | 16 | 20 | 17
  Pain, Grade 3 | 2 | 1 | 1 | 1 | 2
  Redness (mm), Any | 0 | 0 | 0 | 0 | 0
  Redness (mm), Grade 3 | 0 | 0 | 0 | 0 | 0
  Swelling (mm), Any | 0 | 0 | 0 | 1 | 0
  Swelling (mm), Grade 3 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: Duration of Solicited Local Symptoms
Description: Duration was defined as number of days with any grade of local symptoms.
Time Frame: During the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after any vaccine dose
Population: Analysis was performed on the Total Analysis was performed on the Total Vaccinated cohort which included all vaccinated subjects for whom data were available.cohort which included all vaccinated subjects for whom data were available.
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Days
  Pain, Dose 1: number analyzed (Participants) | 11 | 10 | 11 | 13 | 12
  Pain, Dose 1 | 3.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0]
  Pain, Dose 2: number analyzed (Participants) | 11 | 9 | 10 | 8 | 12
  Pain, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.5 [1.0 to 2.0] | 1.0 [1.0 to 2.5]
  Pain, Dose 3: number analyzed (Participants) | 17 | 13 | 10 | 10 | 12
  Pain, Dose 3 | 1.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 2.0]
  Swelling, Dose 1: number analyzed (Participants) | 0 | 0 | 0 | 1 | 0
  Swelling, Dose 1 |  |  |  | 3.0 [3.0 to 3.0] |

17. Secondary Outcome: Number of Subjects Reporting Solicited General Symptoms.
Description: Assessed solicited general symptoms were fever (defined as temperature ≥ 38.0 degrees Celsius (°C) assessed by any route (oral, axillary, rectal)], irritability/fussiness, drowsiness and. loss of appetite. Any = occurrence of the symptom regardless of intensity grade. Grade 3 irritability/Fussiness and Drowsiness = Prevented normal activity, Grade3 Loss of appetite = Did not eat at all. Grade 3 fever = fever > 40.0 °C. Related = symptom assessed by the investigator as related to the vaccination
Time Frame: During the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after any vaccine dose
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Drowsiness, Any | 25 | 18 | 13 | 17 | 16
  Drowsiness, Grade 3 | 2 | 3 | 1 | 1 | 0
  Drowsiness, Related | 22 | 14 | 12 | 13 | 14
  Irritability / Fussiness, Any | 24 | 17 | 19 | 22 | 21
  Irritability / Fussiness, Grade 3 | 3 | 2 | 3 | 2 | 0
  Irritability / Fussiness, Related | 22 | 14 | 17 | 16 | 19
  Loss Of Appetite, Any | 24 | 13 | 14 | 20 | 13
  Loss Of Appetite, Grade 3 | 0 | 1 | 2 | 2 | 0
  Loss Of Appetite, Related | 21 | 7 | 11 | 15 | 10
  Temperature/(Axillary) (°C), Any | 24 | 17 | 14 | 14 | 10
  Temperature/(Axillary) (°C), Grade 3 | 0 | 0 | 1 | 0 | 0
  Temperature/(Axillary) (°C), Related | 22 | 12 | 12 | 14 | 10

18. Secondary Outcome: Duration of Solicited General Symptoms.
Description: Duration was defined as number of days with any grade of general symptoms.
Time Frame: During the 7-day follow-up period (i.e. on the day of vaccination and 6 subsequent days) after any vaccine dose
Population: as for outcome 15
Measure: Median (Inter-Quartile Range); unit: Days
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Days
  Drowsiness, Dose 1: number analyzed (Participants) | 15 | 10 | 7 | 10 | 11
  Drowsiness, Dose 1 | 2.0 [1.0 to 3.0] | 1.5 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 2.0]
  Drowsiness, Dose 2: number analyzed (Participants) | 15 | 12 | 8 | 9 | 6
  Drowsiness, Dose 2 | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 2.5] | 2.0 [2.0 to 3.5] | 2.0 [1.0 to 2.0] | 1.5 [1.0 to 2.0]
  Drowsiness, Dose 3: number analyzed (Participants) | 11 | 7 | 5 | 10 | 7
  Drowsiness, Dose 3 | 2.0 [1.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.0 [2.0 to 2.0] | 2.5 [1.0 to 4.0] | 1.0 [1.0 to 3.0]
  Irritability / fussiness, Dose 1: number analyzed (Participants) | 13 | 9 | 11 | 13 | 12
  Irritability / fussiness, Dose 1 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 2.0]
  Irritability / fussiness, Dose 2: number analyzed (Participants) | 17 | 12 | 12 | 12 | 16
  Irritability / fussiness, Dose 2 | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 4.0] | 2.0 [1.0 to 3.0]
  Irritability / fussiness, Dose 3: number analyzed (Participants) | 8 | 5 | 8 | 10 | 10
  Irritability / fussiness, Dose 3 | 2.0 [2.0 to 3.0] | 3.0 [2.0 to 3.0] | 1.0 [1.0 to 2.0] | 4.0 [3.0 to 5.0] | 1.5 [1.0 to 3.0]
  Loss of appetite, Dose 1: number analyzed (Participants) | 12 | 5 | 9 | 10 | 8
  Loss of appetite, Dose 1 | 2.0 [1.0 to 2.5] | 3.0 [3.0 to 3.0] | 2.0 [1.0 to 3.0] | 2.5 [2.0 to 5.0] | 1.5 [1.0 to 2.5]
  Loss of appetite, Dose 2: number analyzed (Participants) | 14 | 7 | 7 | 9 | 6
  Loss of appetite, Dose 2 | 2.0 [1.0 to 6.0] | 2.0 [1.0 to 2.0] | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0] | 2.0 [1.0 to 3.0]
  Loss of appetite, Dose 3: number analyzed (Participants) | 12 | 4 | 4 | 11 | 5
  Loss of appetite, Dose 3 | 2.0 [1.0 to 3.5] | 2.5 [1.5 to 4.5] | 2.0 [1.5 to 3.0] | 3.0 [2.0 to 4.0] | 2.0 [1.0 to 3.0]
  Temperature, Dose 1: number analyzed (Participants) | 11 | 5 | 3 | 7 | 5
  Temperature, Dose 1 | 1.0 [1.0 to 1.0] | 2.0 [1.0 to 2.0] | 1.0 [1.0 to 2.0] | 2.0 [1.0 to 4.0] | 1.0 [1.0 to 1.0]
  Temperature, Dose 2: number analyzed (Participants) | 18 | 12 | 9 | 8 | 8
  Temperature, Dose 2 | 1.0 [1.0 to 3.0] | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 1.0] | 1.0 [1.0 to 1.5] | 1.0 [1.0 to 1.0]
  Temperature, Dose 3: number analyzed (Participants) | 4 | 4 | 3 | 3 | 0
  Temperature, Dose 3 | 1.0 [1.0 to 1.5] | 2.0 [1.0 to 3.0] | 1.0 [1.0 to 1.0] | 3.0 [2.0 to 4.0] |

19. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs) Post Primary Vaccination.
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any is defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination. Grade 3 AE = an AE which prevents normal, everyday activities. Related = AE assessed by the investigator as related to the vaccination.
Time Frame: During the 21-day follow-up period (Day 0-Day 20) after each vaccine dose
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Any | 21 | 20 | 23 | 20 | 21
  Grade 3 | 3 | 1 | 1 | 3 | 5
  Related | 2 | 0 | 1 | 1 | 3

20. Secondary Outcome: Number of Subjects Reporting Any Unsolicited Adverse Events (AEs) Post Booster Vaccination
Description: as for outcome 19
Time Frame: During the 30-day (Day 385-Day 415) follow-up period after vaccination
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 36 | 34 | 38 | 35 | 33
Participants
  Any | 16 | 8 | 16 | 19 | 14
  Grade 3 | 1 | 0 | 0 | 1 | 0
  Related | 1 | 0 | 1 | 0 | 0

21. Secondary Outcome: Number of Subjects Reporting Medically Attended Events (MAEs)
Description: MAEs are adverse events with medically-attended visits that were not routine visits for physical examination or vaccination. Any MAE was defined as at least 1 MAE experienced.
Time Frame: During the entire study period (Day 0 to Day 415 approximately)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Any | 29 | 28 | 33 | 27 | 26
  Related | 1 | 0 | 0 | 1 | 0

22. Secondary Outcome: Number of Subjects Reporting Potential Immune Mediated Diseases (pIMDs)
Description: Potential immune-mediated diseases (pIMDs) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology. "Any pIMD" = at least one pIMD experienced by the study subject. Related = pIMD assessed by the investigator to be causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 to Day 415 approximately)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Any | 0 | 0 | 1 | 0 | 0
  Related | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events (SAEs)
Description: A serious adverse event was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
Time Frame: During the entire study period (Day 0 to Day 415 approximately)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Any | 5 | 6 | 10 | 4 | 4
  Related | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Subjects Reporting Adverse Events of Special Interest (AESI)
Description: AESI are a subset of adverse events defined in the Committee for Medicinal Products for Human Use (CHMP) Risk Management Plan for Pandemic Vaccines for safety monitoring.
Time Frame: During the entire study period (Day 0 to Day 415 approximately)
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
Number analyzed (Participants) | 38 | 37 | 38 | 37 | 35
Participants
  Any | 4 | 3 | 3 | 2 | 2
  Related | 1 | 0 | 1 | 1 | 0

ADVERSE EVENTS:
Time Frame: Solicited local and general AEs: during 7-day follow-up period after any vaccine dose. Unsolicited AEs: Days 0-20 after each primary dose and Days 385-415 post booster dose . MAEs, pIMDs, SAEs, AESI: during the entire study period (Days 0-415 approximately).
Description: The analysis was performed solely on vaccinated subjects with symptom sheet completed for the reported specific symptom.
Arm/Group | H5N1 Formulation 1 Group | H5N1 Formulation 2 Group | H5N1 Formulation 3 Group | H5N1 Formulation 4 Group | H5N1 Formulation 5 Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/37 | 0/38 | 0/37 | 0/35
Serious Adverse Events (participants affected / at risk) | 5/38 | 6/37 | 10/38 | 4/37 | 4/35
Other Adverse Events (participants affected / at risk) | 36/38 | 31/37 | 35/38 | 35/37 | 32/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H5N1 Formulation 1 Group (N=38) | H5N1 Formulation 2 Group (N=37) | H5N1 Formulation 3 Group (N=38) | H5N1 Formulation 4 Group (N=37) | H5N1 Formulation 5 Group (N=35)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bacteraemia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bacterial infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Croup infectious (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea infectious (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Herpangina (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oral herpes (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 1 (1) | 0 (0)
Pneumonia respiratory syncytial viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Scarlet fever (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tonsillitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Varicella (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Viral rash (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 1 (1) | 1 (1) | 1 (3) | 0 (0) | 0 (0)
Balanoposthitis (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Kawasaki's disease (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | H5N1 Formulation 1 Group (N=38) | H5N1 Formulation 2 Group (N=37) | H5N1 Formulation 3 Group (N=38) | H5N1 Formulation 4 Group (N=37) | H5N1 Formulation 5 Group (N=35)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Acute sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Body height below normal (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body temperature increased (Investigations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 1 (1)
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bronchiolitis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bronchitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 2 (2) | 3 (3) | 1 (2)
Decreased appetite (Metabolism and nutrition disorders) | 25 (39) | 13 (16) | 14 (20) | 20 (30) | 13 (19)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 1 (1) | 2 (2) | 3 (3)
Eczema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterovirus infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Erythema of eyelid (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eyelid oedema (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Failure to thrive (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Febrile convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Feeling hot (General disorders) | 2 (4) | 0 (0) | 3 (3) | 1 (1) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Forearm fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Foreign body in eye (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 2 (3) | 1 (1) | 0 (0) | 0 (0)
Gastroenteritis viral (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hand-foot-and-mouth disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hordeolum (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Impetigo (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Injection site erythema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site urticaria (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 24 (39) | 17 (26) | 19 (31) | 22 (35) | 21 (38)
Limb injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mouth ulceration (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nasopharyngitis (Infections and infestations) | 10 (13) | 8 (10) | 10 (15) | 5 (6) | 9 (10)
Oral herpes (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis media acute (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 20 (39) | 15 (32) | 16 (31) | 20 (31) | 17 (36)
Paronychia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 3 (6) | 1 (1) | 5 (5) | 1 (1) | 3 (3)
Pharyngotonsillitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 24 (36) | 17 (21) | 15 (16) | 16 (20) | 12 (15)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash generalised (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Rash papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiration abnormal (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Respiratory syncytial virus bronchitis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 5 (7) | 1 (3) | 2 (2)
Roseola (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Skin abrasion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Somnolence (Nervous system disorders) | 25 (42) | 18 (29) | 13 (20) | 17 (29) | 16 (24)
Speech disorder developmental (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tonsillitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 7 (7) | 8 (10) | 6 (6) | 13 (16) | 8 (9)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Viral diarrhoea (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Viral rash (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Viral upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 0 (0) | 1 (1) | 2 (2) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.

DOCUMENTS (2):
  • Study Protocol (2017-03-27): https://cdn.clinicaltrials.gov/large-docs/43/NCT02719743/Prot_000.pdf
  • Statistical Analysis Plan (2018-03-01): https://cdn.clinicaltrials.gov/large-docs/43/NCT02719743/SAP_001.pdf